CLINICAL TRIAL: NCT07141251
Title: Multicenter, Open-labeled, Single-arm Clinical Trial of Multi-Branch AOrtic Reconstruction of Complex Aortic Aneurysm With G-iliac System [BAO-G] Technique
Brief Title: Clinical Trial of BAO-G Technique in Complex Aortic Aneurysm Endovascular Repair (BAO-G-02)
Acronym: BAO-G-02
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Fudan University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Changhai Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Beijing Anzhen Hospital (Other); RenJi Hospital (Other); Hainan General Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Jining Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAO-G-02
Record Dates: First submitted 2025-08-11; First posted 2025-08-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Thoracoabdominal Aortic Aneurysm; Endovascular Repair; Complex Aortic Aneurysms
Keywords: BAO-G technique; iliac-branched devices; endovascular repair; complex aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAO-G group (Experimental)
  Interventions: Procedure: BAO-G

INTERVENTIONS:
Procedure: BAO-G — Using G-iliac system to reconstruct the visceral branches of in endovascular repair of thoracoabdominal aortic aneurysm.

SUMMARY:
Multi-Branch AOrtic Reconstruction With G-iliac System (BAO-G) Technique is a novel technique of endovascular repair of complex aortic aneurysm, which using off-the-shelf iliac branched devices to reconstruct the visceral branches. This study aims to verify the perioperative safety and 5-year efficacy of BAO-G technique in the endovascular treatment of complex aortic aneurysms through a prospective, multicenter, open-label, single-arm clinical trial, and to provide evidence for the selection of clinical procedures for complex aortic aneurysm patients in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Crawford type III-IV thoracoabdominal aortic aneurysm or complex abdominal aortic aneurysm, with a healthy proximal landing zone (>20mm length, angulation <60°) in the descending aorta and maximum aneurysm diameter ≥4cm
2. Scheduled for endovascular aortic repair with commercially available iliac branch devices for visceral artery reconstruction
3. Signed informed consent and committed to protocol-defined follow-up

Exclusion Criteria:

1. Acquired language barrier, intellectual decline, cognitive impairment, or mental illness preventing informed consent
2. Uncontrolled autoimmune diseases (e.g., Takayasu arteritis, systemic lupus erythematosus, vasculitis)
3. Prior aortic surgery with stent-graft or prosthetic vascular graft implantation
4. End-stage renal/hepatic/cardiac/pulmonary failure or malignancy diagnosed within 5 years, likely to cause mortality during follow-up
5. Active bleeding or coagulopathy within 6 months (high bleeding risk)
6. Uncontrolled hypertension (resting SBP >180 mmHg or DBP >110 mmHg)
7. Uncontrolled diabetes (fasting blood glucose >16.7 mmol/L)
8. Severe hepatic/renal dysfunction (serum creatinine >3 mg/dL, ALT/AST >3×ULN)
9. Concurrent participation in other interventional clinical trials
10. Pregnancy or perinatal status
11. Refusal to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of primary technical success | within 30 days postoperatively
  The preoperative planned protocol was successfully completed, including aneurysm repair and visceral branch reconstruction, with no aneurysm-related conversion to open surgery/death, no type I/III endoleak, and no branch occlusion within 30 days postoperatively.
Incidence of clinical success | within 5 years postoperatively
  The preoperative planned protocol was successfully completed, including aneurysm repair and visceral branch reconstruction, without significant disabling permanent clinical sequelae, and with the patient remained free from aneurysm-related mortality or secondary interventions due to aneurysm progression during follow-up.

SECONDARY OUTCOMES:
Incidence of aneurysm-related death occurred during perioperative period | within 30 days postoperatively
  All deaths occurring before discharge or within 30 days postoperatively that were attributable to the surgical treatment (including stent-induced retrograde dissection, procedure-related aneurysm rupture, branch occlusion causing severe visceral ischemia, etc.) or aneurysm progression, unless there is clear evidence demonstrating the patient's death was unrelated to the aneurysm.
Incidence of rupture of aneurysms | within 5 years postoperatively
Incidence of permanent paraplegia | within 5 years postoperatively
Incidence of permanent lower limb monoparesis | within 5 years postoperatively
Incidence of new-onset dialysis-dependent renal failure | within 5 years postoperatively
Incidence of severe bowel ischemia | within 5 years postoperatively
Incidence of disabling stroke | within 5 years postoperatively
Intraoperative blood loss | during the operation
Incidence of vascular access complications | within 5 years postoperatively
Operative time | during the operation
Length of stay (LOS) | From the date of hospital admission until the date of hospital discharge, assessed up to 5 years
Length of stay for planned staged procedures | From the date of hospital admission until the date of hospital discharge, assessed up to 5 years
Incidence of adjunctive primary technical success | within 30 days postoperatively
  Required unplanned additional endovascular techniques (e.g., parallel stent-graft technique) to achieve aneurysm exclusion, without type I/III endoleak and with branch patency for 30 days
Incidence of secondary technical success | within 30 days postoperatively
  Required unplanned surgical conversion to complete aneurysm exclusion, without type I/III endoleak and with branch patency for 30 days.
Incidence of stent migration | within 5 years postoperatively
  Definitive stent migration (≥10mm axial displacement) confirmed by evaluation using anatomical landmarks on the first postoperative CT.
Incidence of aneurysm enlargement | within 5 years postoperatively
  Aneurysm enlargement (>5mm maximum diameter increase) demonstrated on perioperative and follow-up CTA.
Incidence of significant distal embolization | within 5 years postoperatively
  Stent-induced lower limb arterial embolism with ischemia requiring surgical intervention, amputation, or resulting in death.
Incidence of Stent- or procedure-related exploratory laparotomy | within 5 years postoperatively
  Adverse event requiring exploratory laparotomy due to stent- or procedure-related complications
Incidence of aortoiliac stent occlusion | within 5 years postoperatively
  Occlusion of aortic branch stents, iliac branch devices, or iliac limb extensions
Rate of primary stent patency | within 5 years postoperatively
  Patency of branch stents and bridging stents, with no in-stent restenosis or occlusion.
Rate of adjunctive primary stent patency | within 5 years postoperatively
  Secondary intervention was required due to branch/bridging stent kinking or in-stent restenosis, with patency restored after the additional procedure.
Rate of secondary stent patency | within 5 years postoperatively
  Patency restored after secondary intervention for branch/bridging stent occlusion.
Incidence of reoperation | within 5 years postoperatively
  Unplanned reoperation related to stent or procedure within the intended treatment zone, excluding access-related reinterventions and procedures outside the target anatomical area.
Incidence of acute kidney injury | within 30 days postoperatively
  A perioperative increase in serum creatinine to 1.5-2 times the preoperative baseline value according to RIFLE criteria.
Incidence of Type I endoleak | within 5 years postoperatively
  Endoleak originating from proximal or distal seal zones
Incidence of Type Ia endoleak | within 5 years postoperatively
  Endoleak originating from the proximal seal zone of aortic stent
Incidence of Type Ib endoleak | within 5 years postoperatively
  Endoleak originating from the distal seal zone of aortic or iliac stents
Incidence of Type Ic endoleak | within 5 years postoperatively
  Endoleak originating from the distal seal zone of visceral artery stents
Incidence of Type II endoleak | within 5 years postoperatively
  Endoleak originating from aortic branches (e.g., inferior mesenteric artery, lumbar arteries, intercostal arteries)
Incidence of Type III endoleak | within 5 years postoperatively
  Endoleak originating from stent junctions or device structural failure
Incidence of Type IIIa endoleak | within 5 years postoperatively
  Endoleak due to aortoiliac stent junctional failure
Incidence of Type IIIb endoleak | within 5 years postoperatively
  Endoleak caused by fracture or disruption of visceral artery stents within branch vessels
Incidence of Type IIIc endoleak | within 5 years postoperatively
  Endoleak into the aortic aneurysm sac due to poor connection or structural failure between visceral branch bridging stents and aortic branch stents
Incidence of Type IV endoleak | within 5 years postoperatively
  Endoleak due to stent-graft fabric permeability

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No